CLINICAL TRIAL: NCT05052736
Title: Effectiveness and Safety of NXsignal Applied Surface Neurostimulation Technology for the Treatment of Type I Complex Regional Pain Syndrome (CRPS I)
Brief Title: Non Invasive Neurostimulation Technology for the Treatment of Type I Complex Regional Pain Syndrome (CRPS I)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Las Palmas de Gran Canaria (Other)
Responsible Party: Principal Investigator, Aníbal Báez Suárez, Principal Investigator, University of Las Palmas de Gran Canaria
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NESAMAZ
Record Dates: First submitted 2021-09-12; First posted 2021-09-22 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Type I Complex Regional Pain Syndrome
Keywords: physical therapy modality; Electric Stimulation Therapy; pain
MeSH Terms: conditions — Reflex Sympathetic Dystrophy; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-invasive Neuromodulation (Experimental): Non-invasive Neuromodulation Intervention with microcurrents: application of 6 electrodes per extremity and an adhesive electrode at C7 level.
  Interventions: Device: Non-invasive Neuromodulation
- Placebo Non-invasive Neuromodulation (Placebo Comparator): Intervention with microcurrents: application of 6 electrodes per extremity and an adhesive electrode at C7.
  Interventions: Device: Non-invasive Neuromodulation

INTERVENTIONS:
Device: Non-invasive Neuromodulation — The electrodes will be placed with the help of gloves and adapted socks for 1 hour, twice a week, until 20 intervention sessions are completed. In addition, depending on the session, an adhesive electrode will be placed at the level of C7.
  Characteristics of microcurrents: pulsed monophasic rectangular wave with a pulse of 1.3 s and pause of 300 ms, voltage 3 millivolt and intensity 0.5 μA.

SUMMARY:
Complex Regional Pain Syndrome (CRPS) / Complex Regional Pain Syndrome (CRPS) is a chronic neurological disorder that affects the extremities and is characterized by disabling pain, swelling, vasomotor instability, sudomotor abnormality, and impaired motor function; the duration and clinical magnitude is greater than expected, being divided into three stages of progression over time: Stage I: acute (0-3 months); Stage II: dystrophic (3-9 months); Stage 3: atrophic (9-18 months).

The purpose of this study is to investigate the effect on complex pain syndrome using a conventional care protocol plus the application of non-invasive neuromodulation during compared to the effect of the same protocol plus placebo.

DETAILED DESCRIPTION:
The design of this study is a randomised, triple blind clinical trial with placebo control.

The size of the sample will be 42 participants who come to referral hospitals. They will be randomized in two groups: control or experimental.

The variables of the study will be collected at three time points: before the intervention, during the intervention and at the end of the intervention.

The variables of the study will be collected at two time points: before the intervention and at the end of the intervention.

The statistical analysis will be an intention-to-treat analysis. For the main outcomes variables a two factor ANOVA will-be performed (intervention-time) with a post-hoc analysis with kruskal wallis correction correction. Statistical significance will be defined as p <0.05

ELIGIBILITY:
Inclusion Criteria:

* Meet the Budapest criteria for the clinical diagnosis of CRPS type I.
* Age between 18 and 65.
* Period between 0 and 6 months after the onset of the clinical picture.
* Have signed the informed consent of their own free will.

Exclusion Criteria:

* Have a diagnosis of CRPS type II.
* Present type I CRPS in more than one limb.
* Patients who have suffered a recurrence of CRPS type I.
* Pregnancy or plans for it during the study.
* Previous sympathectomy in the affected limb.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-03-28 (Actual); Primary Completion 2026-04-27 (Estimated); Study Completion 2026-12-27 (Estimated)

PRIMARY OUTCOMES:
Pain ( VAS) | Up to 6 month
  The instrument will be used to measure the change of pain before and after the intervention will be the Visual Analogue Scale (VAS).
  Participants will be asked to mark the level of their pain on a 100 mm, no hatched VAS scale marked at one end as "no pain" and at the other as "worst pain imaginable".
Quick Dash Test | Up to 6 month
  The Quick DASH Upper Extremity Rating Scale for Upper Extremity can be completed by the patient in aid of the orthopedic surgeon. It consists of 11 items that assess the presence of symptoms and the functional capacity of the individual surveyed during the last week. A total of 11 questions must be answered for the questionnaire to calculate the functional situation accurately

SECONDARY OUTCOMES:
Muscle balance | Up to 6 month
  The Daniels scale or Daniels test is a tool used to measure the strength of muscles in the human body, especially in patients with neuromuscular disorders or localized injuries.
  the scale itself follows a specific numbering, with six well-differentiated levels from 0 to 5. These are the following:
  0: the muscle does not contract, complete paralysis.
  1. the muscle contracts, but there is no movement. The contraction can be palpated or visualized, but there is no movement.
  2. the muscle contracts and performs all the movement, but without resistance, since it cannot overcome gravity.
  3. the muscle can carry out the movement against gravity as the only resistance.
  4. the muscle contracts and performs the full movement, in full range, against gravity and against moderate manual resistance.
  5. the muscle contracts and performs the movement in full range against gravity and with maximum manual resistance
Sleep quality | Up to 6 month
  The Medical Outcomes Study Sleep Scale questionnaire will be used. This instrument was designed to obtain subjective information on the quality and quantity of sleep in the last 4 weeks. It is composed of 12 Likert-type items with 6 degrees of response (from 1-always to 6-never) and grouped into the following categories:
  * Sleep disturbances
  * snoring
  * Waking up with shortness of breath or headache
  * Amount of sleep
  * Adequacy of sleep
  * Daytime sleepiness
  For its interpretation, a gross estimate of the amount of sleep is obtained (item 2) and scores in the different subscales. The direct scores are transformed into a scale from 0 to 100, with no cut-off points; the higher the score, the greater the intensity of the concept evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Aníbal Báez-Suárez, PhD, Principal Investigator — University of Las Palmas de Gran Canaria
Locations (1):
- Aníbal Báez Suárez, Las Palmas de Gran Canaria, Palmas, Las, Spain

REFERENCES:
- [Result] Sebastin SJ. Complex regional pain syndrome. Indian J Plast Surg. 2011 May;44(2):298-307. doi: 10.4103/0970-0358.85351. PMID 22022040
- [Result] Wasner G, Schattschneider J, Binder A, Baron R. Complex regional pain syndrome--diagnostic, mechanisms, CNS involvement and therapy. Spinal Cord. 2003 Feb;41(2):61-75. doi: 10.1038/sj.sc.3101404. PMID 12595868
- [Result] Todorova J, Dantchev N, Petrova G. Complex regional pain syndrome acceptance and the alternative denominations in the medical literature. Med Princ Pract. 2013;22(3):295-300. doi: 10.1159/000343905. Epub 2012 Nov 16. PMID 23171669
- [Result] Bruehl S. An update on the pathophysiology of complex regional pain syndrome. Anesthesiology. 2010 Sep;113(3):713-25. doi: 10.1097/ALN.0b013e3181e3db38. PMID 20693883
- [Result] Ratti C, Nordio A, Resmini G, Murena L. Post-traumatic complex regional pain syndrome: clinical features and epidemiology. Clin Cases Miner Bone Metab. 2015 Jan-Apr;12(Suppl 1):11-6. doi: 10.11138/ccmbm/2015.12.3s.011. Epub 2016 Apr 7. PMID 27134626
- [Result] Sandroni P, Benrud-Larson LM, McClelland RL, Low PA. Complex regional pain syndrome type I: incidence and prevalence in Olmsted county, a population-based study. Pain. 2003 May;103(1-2):199-207. doi: 10.1016/s0304-3959(03)00065-4. PMID 12749974
- [Result] Elsamadicy AA, Yang S, Sergesketter AR, Ashraf B, Charalambous L, Kemeny H, Ejikeme T, Ren X, Pagadala P, Parente B, Xie J, Lad SP. Prevalence and Cost Analysis of Complex Regional Pain Syndrome (CRPS): A Role for Neuromodulation. Neuromodulation. 2018 Jul;21(5):423-430. doi: 10.1111/ner.12691. Epub 2017 Sep 29. PMID 28961359
- [Result] Albazaz R, Wong YT, Homer-Vanniasinkam S. Complex regional pain syndrome: a review. Ann Vasc Surg. 2008 Mar;22(2):297-306. doi: 10.1016/j.avsg.2007.10.006. PMID 18346583